CLINICAL TRIAL: NCT02857933
Title: Daily and Weekly Rehabilitation Delivery for Young Children With Gross Motor Delays
Acronym: DRIVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jill Heathcock, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015N0054
Record Dates: First submitted 2016-06-22; First posted 2016-08-05 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Gross Motor Development Delay
Keywords: Motor Impairments; Gross Motor Delay
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Frequency Level 1 - Daily Therapy (Other): Level 1 daily physical therapy is 2 hours of one-on-one physical therapy per day for 20 straight weekdays
  Interventions: Other: Physical Therapy
- Frequency Level 2 - Intermediate Therapy (Other): Level 2 intermediate physical therapy is 2 hours of therapy per day 3 days per week for 6.6 weeks
  Interventions: Other: Physical Therapy
- Frequency Level 3 - Usual Therapy (Other): Level 3 usual weekly physical therapy is 2 hours of therapy one day per week for 20 weeks.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — One-on-one physical therapy sessions (one therapist and one patient). Principles of motor learning used include repetition, task-specificity, active practice, generalization of skills, errors, structured practice, and developmentally appropriate feedback with sufficient time to practice.

SUMMARY:
The purpose of this study is to determine the optimal frequency and intensity of physical therapy for children with cerebral palsy aged 6 to 24 months of age. Participants will be randomly assigned to one of three groups: daily, intermediate, or weekly physical therapy. Short and long term effects will be evaluated to determine the best 'dose' of rehabilitation for children with cerebral palsy, including frequency (number of sessions per week and the number of weeks), intensity (how hard the patient works), and time (how many total hours) of rehabilitation treatment.

DETAILED DESCRIPTION:
Determining optimal frequency of treatment for young children with cerebral palsy (CP) has implications for shaping the future of pediatric rehabilitation. There are wide variations in the number of hours per week of treatment in current outpatient rehabilitation programs for children with CP, suggesting clinical uncertainty. Usual weekly therapy at 1 - 2 hours per week for 6 months or longer is the most commonly implemented frequency of dose for children with CP 6 - 24 months of age. However, this decision about frequency is often made based on clinical reasoning and scheduling, not on principles of rehabilitation, child development, or evidence from strongly designed randomized controlled trials. The proposed study will fill this gap by directly comparing the effects of 3 frequency levels of therapy - concentrated daily, intermediate, and usual weekly in children with CP 6 - 24 months of age at the initiation of treatment and following these patients for 2 years.

In this prospective longitudinal study, children with Cerebral Palsy (n=75), 6 - 24 months of age, will be randomly assigned to one of three groups: daily, intermediate, or weekly physical therapy. The treatment phase of this study design is 5 months for a total of 40 hours of one-on-one therapy for both groups. Level 1 daily therapy is 2 hours of therapy per day for 20 straight weekdays. Level 2 intermediate therapy is 2 hours of therapy per day 3 days per week for 6.6 weeks. Level 3 usual weekly therapy is 2 hours of therapy one day per week for 20 weeks. Researchers will directly compare the effects of 3 these frequency levels of therapy at the initiation of treatment and following these patients for 2 years. Results will provide quantitative evidence of frequency-response, which is critical for informing clinical decision-making, health policy, and guidelines for reimbursement.

ELIGIBILITY:
Inclusion Criteria:

* an age of 6 months - 24 months at the initiation of treatment. The age will be corrected for any eligible children born preterm until they are 2 years of age, as is standard clinical and research practice
* a diagnosis or risk for CP in GMFCS levels III, IV and V or motor delay
* ability to tolerate a 2 hour therapy session based on parent report and evaluating therapists, the same criteria the investigators used for the pilot study.

Exclusion Criteria:

* uncontrollable seizures or any co-morbid condition that prevents full participation during treatment sessions
* participation in another daily treatment program in the last 6 months
* auditory, or visual conditions that prevent full participation during treatment sessions
* progressive neurological disorder with no potential for improvement.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2024-10 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure (GMFM)-88 | Baseline (pre-treatment) and 3 months, 6 months, 12 months, 18 months, and 24 months after initiation of treatment
  GMFM evaluates change in gross motor function over time or with intervention in children with CP from 5 months to 16 years. It has been used widely in the field to determine functional motor change following intervention.

SECONDARY OUTCOMES:
Change in Goal Attainment Scaling (GAS) | Baseline (pre-treatment) and 3 months, 6 months, 12 months, 18 months, and 24 months after initiation of treatment
  GAS creates patient, family, and clinical anchors as the external criterion for improvement by establishing activity or participation goals that reflect what an individual, family, and clinician consider meaningful or relevant.The GAS method allows for goals to be defined at different levels of mastery and assigned numerical values for score calculation, similar to a Likert scale. The scale will have 5 points representing different levels of mastery of the individual patient's goal. A score of -2 represents baseline, -1 less change than expected, 0 for the expected level of change, and +1 and +2 for achievement of more change than expected. To attempt to ensure ordinality, each level on the scale will be described and will reflect a single dimension of change that is measureable, achievable, and relevant
Change in Bayley Scales of Infant Development III | Baseline (pre-treatment) and 3 months, 6 months, 12 months, 18 months, and 24 months after initiation of treatment
  The Bayley Scales of Infant and Toddler Development-Third Edition is an individually administered test designed to assess developmental functioning of infants and toddlers. The Bayley-III assesses development in five areas: cognitive, language, motor, social-emotional, and adaptive behavior.
Change in Pediatric Evaluation and Disability Inventory (PEDI) | Baseline (pre-treatment) and 3 months, 6 months, 12 months, 18 months, and 24 months after initiation of treatment
  Administered as a parent survey. The PEDI is a descriptive measure of a child's current functional performance and can track changes over time. The PEDI measures both capability and performance of functional activities in three content domains: self-care, mobility, and social function.It can be used as a comprehensive clinical assessment of key functional capabilities and performance in children between the ages of six months and seven years.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Heathcock, MPT, PhD, Principal Investigator — Ohio State University
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Scott K, Lewis J, Pan X, Heathcock J. Parent-Reported PEDI-CAT Mobility and Gross Motor Function in Infants With Cerebral Palsy. Pediatr Phys Ther. 2021 Jul 1;33(3):156-161. doi: 10.1097/PEP.0000000000000801. PMID 34086623
- [Derived] Ferrante R, Hendershot S, Baranet K, Barbosa G, Carey H, Maitre N, Lo W, Pan J, Heathcock J. Daily and Weekly Rehabilitation Delivery for Young Children With Gross Motor Delay: A Randomized Clinical Trial Protocol (the DRIVE Study). Pediatr Phys Ther. 2019 Apr;31(2):217-224. doi: 10.1097/PEP.0000000000000594. PMID 30865149